CLINICAL TRIAL: NCT00003253
Title: Assessment of the Predictive Value of the Extreme Drug Resistance (EDR) Assay in Patients Receiving Paclitaxel for Metastatic Breast Cancer
Brief Title: Evaluation of Drug Resistance in Patients With Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oncotech (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: CDR0000066135; ONCOTECH-OTBR01; UCIRVINE-97-02; NCI-V98-1391
Record Dates: First submitted 1999-11-01; First posted 2003-11-26 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2006-05

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Paclitaxel; Drug Screening Assays, Antitumor

INTERVENTIONS:
Drug: paclitaxel
Other: antitumor drug screening assay

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Some patients may develop a resistance to chemotherapy drugs.

PURPOSE: Phase II trial to determine the reliability of a test for measuring drug resistance to paclitaxel in patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the proportion of patients with extreme, intermediate, and low drug resistance to paclitaxel using the Extreme Drug Resistance (EDR) Assay in patients with previously treated metastatic breast cancer. II. Assess response to paclitaxel therapy in patients who have undergone a pretreatment EDR assay. III. Assess time to tumor progression during paclitaxel therapy in patients who have undergone a pretreatment EDR assay. IV. Determine prospectively the predictive value of the EDR assay relative to clinical outcome by correlating assay results with clinical tumor response and time to tumor progression during paclitaxel therapy in these patients.

OUTLINE: This is an open label, single arm, blinded study. Patients' tumor tissue samples are collected by excisional biopsy, core biopsy, or malignant fluid aspiration, then tested by the Extreme Drug Resistance (EDR) Assay to determine probability of drug resistance to paclitaxel. After successful completion of the EDR assay (approximately 7 days), patients receive paclitaxel by intravenous infusion over 1-3 hours; treatment is repeated every 3 weeks. Treatment continues until there is documented evidence of tumor progression or unacceptable toxicity. Patients' clinical response to paclitaxel therapy is compared with the response predicted by the EDR assay.

PROJECTED ACCRUAL: 100 patients will be accrued to this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Metastatic breast cancer that is accessible for biopsy or aspiration Bidimensionally measurable disease with at least one diameter greater than 1 cm documented on x-ray or photograph, or a palpable lesion No brain metastases or carcinomatous meningitis Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Male or female Menopausal status: Not specified Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT no greater than 3 times upper limit of normal (ULN) (no greater than 5 times ULN if metastatic to liver) Renal: Creatinine no greater than 2.0 mg/dL Calcium no greater than 12 mg/dL Cardiovascular: No myocardial infarction within 3 months prior to study No unstable angina or symptomatic congestive heart failure Other: No active or uncontrolled infection Not HIV positive No psychoses Not pregnant or nursing Effective contraception required of fertile women No second malignancy within past 5 years except: Adequately treated basal or squamous cell carcinoma of the skin In situ cancer of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Prior paclitaxel permitted if patient had disease-free interval of greater than 1 year Prior taxotere permitted Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 1997-07

CONTACTS AND LOCATIONS:
Overall Officials: Rita S. Mehta, MD, Study Chair — Oncotech
Locations (9):
- United States (9):
  - Pacific Coast Hematology/Oncology Medical Group, Fountain Valley, California
  - Long Beach Memorial Breast Center, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Howard University, Washington D.C., District of Columbia
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Palmetto Hematology/Oncology Associates, Spartanburg, South Carolina
  - University of Texas - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Fruehauf JP, Mehta RS, Parker RJ: Association of invitro resistance to paclitaxel with clinical outcome in metastatic breast cancer patients with taxol: a multi-institutional prospective trial. [Abstract] Proc Am Assoc Cancer Res 41: A-2096, 330, 2000.